CLINICAL TRIAL: NCT04169022
Title: Targeting Interleukin 1 Receptor Accessory Protein (IL1RAP) Expressing Acute Myeloid Leukemic (AML) Cells by Chimeric Antigen Receptor (CAR) Engineered T-cells
Brief Title: AML Cell Immunotherapy Using Chimeric Antigen Receptor T-cells
Acronym: CAR-LAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: P/2018/402
Record Dates: First submitted 2019-05-16; First posted 2019-11-19 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Chimeric Antigen Receptor T Cells; Immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AML patients at diagnosis (Experimental): AML patients at diagnosis (except AML3)
  Interventions: Other: Sample collection
- AML patients at relapse (Experimental): AML patients at relapse after chemotherapy, targeted therapy or allograft
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — Sample collection blood and/or bone marrow

SUMMARY:
AML is one of the most aggressive forms of leukemia, where bone marrow transplantation remains the gold standard treatment, with its known associated toxicities and related mortality. Despite progress in the treatment of leukemic malignancies, especially the emergence of targeted- and immuno-therapies arising from biological genomic knowledge, there remains a need to provide additional strategies for refractory/relapsing (R/R) patients

Aim of this study is to collect biological samples of AML patients in order to validate our Chimeric Antigen Receptor T-cells immunotherapy approach

ELIGIBILITY:
Inclusion Criteria:

* AML patients adults and pediatrics

Exclusion Criteria:

* AML3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
IL1RAP protein expression | 2 years
  Cytometry analysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, France